CLINICAL TRIAL: NCT06094101
Title: Prospective Phase I/II Trial of an Individualized Peptide Vaccine in Pediatric and AYA Patients with Metastasized Fusion-driven Sarcomas Following Standard Treatment
Brief Title: Personalized Vaccination in Fusion+ Sarcoma Patients (PerVision)
Acronym: PerVision
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Deutsches Konsortium fürTranslationale Krebsforschung (DKTK) (Unknown); Cooperative Ewing Sarkom Studiengruppe (Unknown); Cooperative Weichteilsarkom Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-002793-91
Record Dates: First submitted 2023-09-25; First posted 2023-10-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Ewing Sarcoma; Rhabdomyosarcoma; Synovial Sarcoma
Keywords: metastasized fusion-driven sarcoma; clinical study; phase I/II
MeSH Terms: conditions — Sarcoma, Ewing; Rhabdomyosarcoma; Sarcoma, Synovial

STUDY DESIGN:
Intervention Model Description: interventional, multicenter, open-label, phase I/II feasibility and early proof of concept study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peptide vaccination (Experimental): Peptides will be administered subcutaneously (s.c.) together with the novel toll like receptor (TLR) 1/2 ligand XS15 emulsified in Montanide ISA 51 VG as adjuvant.
  Three vaccinations will be applied every 28 days.
  Interventions: Biological: Peptide vaccine IPX

INTERVENTIONS:
Biological: Peptide vaccine IPX — Peptide vaccine is a combination of
  1. class II peptide spanning the sarcoma-specific fusion-breakpoint (fusion-peptide)
  2. class-II neopeptide based on a patient-individual nonsynonymous mutation with a high immunogenicity (mutation-based neopeptide).
  3. control peptide derived from Survivin.
  4. adjuvant: toll like receptor (TLR) 1/2 ligand XS15.

SUMMARY:
The PerVision trial utilizes an approach of a patient-individual cancer vaccine with sarcoma-specific peptides in metastasized fusion-driven sarcoma patients determined by next generation whole exome sequencing of tumor and normal tissue as well as RNA sequencing of the tumor.

This approach is applicable to all patients independent of the expression of distinct tumor associated antigens, and independent of their human leukocyte antigen-typing (HLA-typing). The results of this study can directly be translated to other tumor entities.

It is an interventional, multicenter, open-label, phase I/II feasibility and early proof of concept study evaluating a personalized peptide vaccine.

Primary objective is to evaluate safety and success of treatment, the latter be defined as vaccination-induced T-cell response without unacceptable toxicity.

DETAILED DESCRIPTION:
The PerVision trial utilizes an approach of a patient-individual cancer vaccine with sarcoma-specific peptides (one peptide derived from the sarcoma-specific fusion breakpoint, 'fusion-peptide', and a second peptide derived from neoantigens derived from patient-specific non-synonymous mutations with the highest prediction score, 'mutation-based neopeptide') in metastasized fusion-driven sarcoma patients determined by next generation whole exome sequencing of tumor and normal tissue as well as RNA sequencing of the tumor.

This approach is applicable to all patients independent of the expression of distinct tumor associated antigens, and independent of their human leukocyte antigen-typing (HLA-typing). The results of this study can directly be translated to other tumor entities.

It is an interventional, multicenter, open-label, phase I/II feasibility and early proof of concept study evaluating a personalized peptide vaccine and the toll like receptor (TLR) 1/2 ligand XS15 emulsified in Montanide ISA 51 VG in fusion driven sarcoma patients.

The principal questions are:

1. To investigate, whether it is possible to induce a mutation-specific immune response in sarcoma patients and young adults after salvage chemotherapy
2. To investigate possible side effects and toxicity of the treatment
3. To gather indications if our approach has a beneficial effect on residual disease as well as event free survival (EFS) of the patients. EFS and overall survival (OS) data will be compared within this single arm study to non-vaccinated patients of a historic control cohort.

Patients will be recruited through the Society for Pediatric Oncology/Hematology (GPOH) networks Cooperative Soft Tissue Sarcoma Group (CWS) and Cooperative Ewing Sarcoma Group (CESS) and through the "Deutsches Konsortium für Translationale Krebsforschung" (DKTK) programs MASTER and INFORM as well as HEROES-AYA. For the screening phase, n=30 patients will be recruited, n=23 patients should be treated with at least one vaccine dose, with a drop-out rate we need n=21 patients for sufficient statistical power.

Primary objective is to evaluate the safety, toxicity and in vivo immunological effects of a patient-individualized peptide vaccination (IPX vaccine) in patients with primary or relapsed metastasized fusion-driven sarcoma (FDS, rhabdomyosarcoma, Ewing- and synovial sarcoma) with an age ≥ 2 to < 40 years in first or second complete remission or stable partial remission.

Primary endpoint is "success of treatment", defined as the patient showing a vaccination-induced T cell response without unacceptable toxicity until Follow-up visit (28 ± 7 days after last vaccination).

ELIGIBILITY:
Inclusion Criteria, definition of partial remission plus (PRplus)

* Screening Stage 1:

  * Confirmed metastatic fusion-driven rhabdomyosarcoma, Ewing- and synovial sarcoma in first or second complete remission (CR) or partial response (PR) after local therapy and intensive standard chemotherapy protocols.
  * Whole exome sequencing and RNA sequencing data of the gene fusion (fusion-breakpoint RNA sequence) must be available by registration to the INFORM (Individualized therapy for relapsed malignancies in childhood), MASTER (Register study Molecularly Aided Stratification for Tumor Eradication) or HEROES-AYA networks (Heterogeneity, evolution and resistance of fusion-driven sarcomas in AYA) or similar evaluation.
* Screening stage 2:

  * Design and production of the patient-individual vaccine cocktail was successful
  * Patients have reached a complete or stable partial remission (CR or PR) the end of adjuvant and/or maintenance cytotoxic treatment. Cytotoxic treatment as per standard or trial recommendations has been completed. Definition of PRplus: Partial remission(plus) implicates that all remaining tumor residua including all metastases have received local therapy by this time point: Either surgical removal or local irradiation. The assessment of which therapy modality and, in the case of irradiation, which radiation dose is selected, lies with the treating physician. Whether PRplus is achieved will be decided finally by the investigator after review of the patient records.

Exclusion Criteria:

* Ejection fraction < 25%
* Creatinine-clearance < 40ml/min
* Bilirubin > 4mg/dl
* Alanine aminotransferase (ALT) > 400 units (U)/l and/or aspartate aminotransferase (AST) > 400 U/l
* Severe infection (Human immunodeficiency virus (HIV): positive for the presence of human immunodeficiency virus-1 or human immunodeficiency virus-2 (positive antigen/antibody or nucleic acid tests [NAT]) and CD4-positive cells < 500/μl. Hepatitis B virus: positive for the presence of hepatitis B virus (positive for hepatitis B core antibody [HBcAb] or positive hepatitis B surface antigen [HBsAg]) and hepatitis B NAT test > 2000 IU/ml). Hepatitis C virus: positive for heavy chain only antibody [HCAb] or for nucleic acid amplification testing (NAT). Other infections that, in the opinion of the investigator, do not allow a participation in the study.)
* Subjects with a known hypersensitivity / allergy to any component of the study drugs.
* Subjects who have received a live, attenuated vaccine within 28 days prior to the administration of the study drug (only stage 2).
* Subjects with a prior haematopoietic stem cell transplantation / prior organ transplantation.
* Patients suffering from other malignancies (with the exception of those with a negligible risk of metastasis or death and treated with curative outcome) within 5 years prior to study start.
* Current or anticipated need for any of the following medications interfering with T cell function from 14 days before 1st vaccination until 28 days after 1st vaccination: Immunosuppressive agents, which influence functionality and activity of T cells, such as steroids (more than 0,5 mg/kg body weight prednisolone-equivalent), calcineurin-inhibitors, mofetil mycophenolate, sirolimus, everolimus, and cytotoxic medication. Those drugs should be avoided until 28 days after third/final vaccination but may be given after discussion with the principal investigator. Application of tyrosine kinase inhibitors is permitted during the trial (only stage 2).
* Significant psychiatric disabilities that, in the judgment of the investigator, do not assure reliable participation in the present study.
* Uncontrolled seizure disorders (occurrence of at least one generalized seizure in the last 3 months) or severe peripheral neuropathy/leucoencephalopathy (> grade 2 according to NCI CTCAE v5.0 neurotoxicity criteria).
* Autoimmune disease (e.g. idiopathic thrombocytopenic purpura, autoimmune hemolytic anemia, autoimmune dermatitis) requiring immunosuppressive treatment
* Pregnant females
* Female subjects of childbearing potential (postmenarcheal, with an intact uterus and at least one ovary, and less than one year postmenopausal) not agreeing to use acceptable method(s) of contraception from 30 days prior to Screening stage 2 visit to 180 days after the last vaccination.
* Male subjects of reproductive capacity not agreeing to use effective contraception from first vaccination of this study to 180 days after the last vaccination.
* Not willing and/or not able to comply with treatment plan, scheduled visits, laboratory tests, contraceptive guidelines and other study procedures.
* History of any illness or clinical condition that might confound the results of the study or pose an additional risk in administering study drug to the subject, according to the judgement of the investigator. This may include but is not limited to: history of central nervous system or cardiovascular disease, history of relevant drug allergies, history of psychiatric disorder, history or present of clinically significant pathology.
* Karnofsky performance status of < 70% for subjects ≥ 16 years of age, Lansky performance status of < 70% for subjects < 16 years of age
* Participation or intended participation in another clinical phase I or II trial with an investigational drug or product within 28 days prior to enrollment (with the exception to participation of the "frontline and relapsed rhabdomyosarcoma study"( (FaR-RMS) after completion of the maintenance therapy (EudraCT-2018-000515-24)). Commonly used drugs as per standard or phase III-trials are permitted.

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Success of treatment | Follow-up visit at 28 +/- 7 days after last vaccination
  The primary composite safety/efficacy outcome of "treatment success" is defined as number of patients
  1. without unacceptable toxicity (any toxicity > grade 3 according to NCI-CTC) until Follow-up visit (28 ± 7 days after last vaccination) and
  2. with vaccination-induced response of cluster of differentiation 4+ (CD4+) and/or cluster of differentiation 8+ (CD8+) T cells to the patient-specific peptides at Follow-up visit (28 ± 7 days after last vaccination). CD4+ and CD8+ T cells will be measured by flow cytometry.

SECONDARY OUTCOMES:
T-cell response at follow up | Beginning of trial phase until follow-up visit at 28 +/- 7 days after last vaccination
  Number of patients with CD8+ and/or CD4+ T-cell responses measured 2-fold above background in response to either of the two patient-specific peptides (fusion-peptide and mutation-based neopeptide).
T-cell response at final follow up | Beginning of trial phase until final follow-up at 120 +/- 14 days after last vaccination
  Number of patients with CD8+ and/or CD4+ T-cell responses measured 2-fold above background in response to either of the two patient-specific peptides (fusion-peptide and mutation-based neopeptide).
Event free survival | Beginning of trial phase until final follow-up at 120 +/- 14 days after last vaccination
  Rate of patients that survived without progression according to RECIST criteria, stratified for immune response yes/no
Overall survival | Beginning of trial phase until final follow-up at 120 +/- 14 days after last vaccination
  Rate of patients that survived. stratified for immune response yes/no
Quality of life (QoL) defined as overall quality of life in children | Beginning of trial phase until final follow-up at 120 +/- 14 days after last vaccination
  QoL (Quality of life) is defined as overall quality of life measured by Pediatric Quality of Life InventoryTM PedsQL (4.0). The PedsQL uses a 0 to 4 scale with 0=never and 4=almost always.
Quality of life (QoL) defined as overall quality of life in adults | Beginning of trial phase until final follow-up at 120 +/- 14 days after last vaccination
  QoL (Quality of life) is defined as overall quality of life measured by European Organisation for Research and Treatment of Cancer EORTC quality of life questionnaire (QLQ) C-30 (3.0). EORTC QLQ C-30 uses a 1-4 scale with 1=not at all and 4=very much and a 1-7 scale with 1=very poor and 7=excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Ebinger, Prof. Dr., Principal Investigator — University children's hospital Tübingen
Locations (4):
- Germany (4):
  - Pediatrics III, West German Cancer Centre, University Hospital, Essen
  - Universitätsklinikum, Klinik für Kinder- und Jugendmedizin, Frankfurt am Main
  - Zentrum für Kinder- und Jugendmedizin, Universitätsklinikum, Freiburg im Breisgau
  - University Children's Hostpital, Tübingen

IPD SHARING:
Plan to Share IPD: No